CLINICAL TRIAL: NCT00969345
Title: Effects of Respiratory Yoga Training (Bhastrika) on Heart Rate Variability and Baroreflex, and Quality of Life of Healthy Elderly Subjects
Brief Title: Effects of Respiratory Yoga Training on Heart Rate Variability and Baroreflex of Healthy Elderly Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Geraldo Lorenzi-Filho, Heart Institute InCor - University of Sao Paulo Medical School
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RESP-HRV
Record Dates: First submitted 2009-08-31; First posted 2009-09-01 (Estimated); Last update posted 2009-09-01 (Estimated); Status verified 2009-08

CONDITIONS: Elderly Subjects; Respiration Exercises
Keywords: Healthy Elderly Subjects; Respiratory Yoga Exercises; Heart Rate Variability; Baroreflex; Quality of Life
MeSH Terms: interventions — Muscle Stretching Exercises

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (Sham Comparator): Stretching exercises performed twice a day for 10 minutes (4 months)
  Interventions: Other: Stretching Exercises
- Respiration Group (Active Comparator): Respiratory Yoga exercises performed twice a day for 10 minutes (4 months)
  Interventions: Other: Respiratory Exercises conducted twice a day for 10 minutes

INTERVENTIONS:
Other: Stretching Exercises — Conducted twice a week, with instructions for home exercises twice a day, and registering each session on a log sheet.
  Arms: Control Group
Other: Respiratory Exercises conducted twice a day for 10 minutes — Conducted twice a week, with instructions for home exercises twice a day, and registering each session on a log sheet.
  Arms: Respiration Group

SUMMARY:
The decreases of physiological capacities which take place with senescence include diminishing respiratory capacity as well as a reduction of heart rate variability and baroreflex sensibility. Altogether, these alterations increase elderly people's frailty and have a negative impact over quality of life. Since Yoga (Indian auto-discipline) has a wide range of respiratory exercises already investigated as components for non-pharmacological treatments for hypertension (situation in which heart rate variability is also diminished), the investigators hypothesis is that the training of respiratory exercises of Yoga may have a significant positive effect on heart rate variability and baroreflex of health elderly subjects, increasing quality of life and reducing frailty.

We included 30 health elderly subjects (both sexes, from 60 years-old onwards) divided into 2 randomized experimental groups: control (C) and respiration (R). Each group underwent an entry evaluation, followed by a 4-months training period, after which they were re-evaluated. Control consisted of 2 stretching classes per week, and respiration consisted of 2 respiratory exercises classes a week. Both groups were instructed to perform the exercises at home twice a day, and to keep a record of each session in a log sheet. Evaluations were: WHOQOL-OLD questionnaire for quality of life, 20 minutes of seated rest with heart rate, respiration and blood pressure acquired continuously for further spectral analysis.

DETAILED DESCRIPTION:
Heart rate variability was performed using the autoregressive model, and the baroreflex was calculated with the spontaneous approach, both with the softwares developed in Milan by Alberto Porta in a non-invasive way.

The frequency domain analysis of heart rate, respiration and systolic blood pressure were conducted, consisting of calculating the power spectral density with the minimum error predicted by Akaike's algorithm. Spectral power was then subdivided into two bands of physiological interest: low - (LF 0.03-0.15 Hz) indicating predominant sympathetic modulation, and high - (HF 0.15-0.5 Hz) frequency, indicating parasympathetic modulation of the heart. The fraction calculated dividing LF by HF (LF/HF ratio) provided information of sympathovagal balance to the heart. The spectral analysis of Systolic Blood Pressure provided information of the vasomotor tone, and the integration of heart rate information with these data also provided information about the spontaneous baroreflex gain.

Other questionnaires used were: Pittsburgh Quality of Sleep Questionnaire, Stress Symptoms Questionnaire by Marilda Lipp - validated in Brazil, and Beck's anxiety and depression inventories.

ELIGIBILITY:
Inclusion Criteria:

* Health elderly subjects

Exclusion Criteria:

* Use of beta-blockers
* Atrial Fibrillation
* Previous training in respiratory exercises

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-08; Primary Completion 2008-07 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Heart Rate Variability | 4 months

SECONDARY OUTCOMES:
baroreflex gain | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Danilo F Santaella, Principal Investigator — Heart Institute (InCor); Geraldo Lorenzi-Filho, MD, PhD, Principal Investigator — Heart Institute
Locations (1):
- Heart Institute (InCor), São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Santaella DF, Devesa CR, Rojo MR, Amato MB, Drager LF, Casali KR, Montano N, Lorenzi-Filho G. Yoga respiratory training improves respiratory function and cardiac sympathovagal balance in elderly subjects: a randomised controlled trial. BMJ Open. 2011 May 24;1(1):e000085. doi: 10.1136/bmjopen-2011-000085. PMID 22021757